CLINICAL TRIAL: NCT00618150
Title: Patient Education in Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Jorgen Urnes/ principal researcher, Norwegian University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Sak 33-96 (REK); SLKNR 96/00515
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; Dyspepsia; Education; Information
MeSH Terms: conditions — Gastroesophageal Reflux; Dyspepsia | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Behavioral: Patient education

INTERVENTIONS:
Behavioral: Patient education — An educational program: Three lessons spaced over 2 weeks.

SUMMARY:
Patients with gastroesophageal reflux disease (heart-burn, acid regurgitation)may benefit from an educational program explaining the medical aspects of the disease, self-management strategies and how to deal with health services. We hypothesized that patients having participated in an educational program would experience an improved quality of life when compared to patients who did not take part (controls).

ELIGIBILITY:
Inclusion Criteria:

* heartburn and acid regurgitation the dominant symptom
* needing relief at least 5 days/ week when symptoms were at their worst
* disease history at least 3 months
* ability to give informed consent

Exclusion Criteria:

* current or previous esophagitis stage 2(Savary-Miller) or greater or peptic ulc
* continuous need of proton pump inhibitors or NSAIDs
* wish for surgical treatment
* earlier surgical treatment in the GI-tract
* pregnancy
* alcohol or drug abuse

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 1996-09; Primary Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Quality of life | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jorgen A Urnes, MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Med. fac., Trondheim, Norway

REFERENCES:
- [Result] Urnes J, Farup PG, Lydersen S, Petersen H. Patient education in gastro-oesophageal reflux disease: a randomized controlled trial. Eur J Gastroenterol Hepatol. 2007 Dec;19(12):1104-10. doi: 10.1097/MEG.0b013e3282f163dc. PMID 17998836
- [Derived] Urnes J, Petersen H, Farup PG. Disease knowledge after an educational program in patients with GERD--a randomized controlled trial. BMC Health Serv Res. 2008 Nov 13;8:236. doi: 10.1186/1472-6963-8-236. PMID 19014552